CLINICAL TRIAL: NCT01163396
Title: Open-label, Multicenter, Phase II Study Of First-line Biweekly Irinotecan, Oxaliplatin And Infusional 5-FU/LV (FOLFOXIRI) In Combination With Bevacizumab In Patients With Metastatic Colorectal Cancer
Brief Title: First-line FOLFOXIRI In Combination With Bevacizumab For Metastatic Colorectal Cancer
Acronym: FOIB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASL606LIOM01
Record Dates: First submitted 2010-07-09; First posted 2010-07-15 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Bevacizumab; Irinotecan; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFOXIRI plus bevacizumab (Experimental): BEVACIZUMAB 5 mg/Kg i.v. followed by IRINOTECAN 165 mg/sqm i.v. over 1 hr followed by OXALIPLATIN 85 mg/sqm i.v. over 2 hr concomitantly with l-LV 200 mg/sqm over 2 hrs followed by 5FU 3.200 mg/sqm c.i. over 48 hrs starting on day 1. Cycles repeated every 2 weeks
  Interventions: Drug: Bevacizumab; Drug: Irinotecan; Drug: Oxaliplatin; Drug: 5-fluorouracil/leucovorin

INTERVENTIONS:
Drug: Bevacizumab
Drug: Irinotecan
Drug: Oxaliplatin
Drug: 5-fluorouracil/leucovorin

SUMMARY:
This is a single-arm, open-label, multicentre phase II study evaluating the safety and efficacy of the combination of the G.O.N.O. FOLFOXIRI regimen with bevacizumab as first-line treatment of metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma
* Unresectable and measurable metastatic disease (RECIST criteria)
* Male or female, aged > 18 years and ≤ 75 years
* ECOG Performance Status (PS) < 2 if aged < 71 years
* ECOG PS = 0 if aged 71-75 years
* Life expectancy of more than 3 months
* Adequate haematological function: ANC ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L, Hb ≥ 9 g/dL
* INR ≤ 1.5 and aPTT ≤ 1.5 x ULN within 7 days prior to starting study treatment
* Adequate liver function: serum bilirubin ≤ 1.5 x ULN; alkaline phosphatase and transaminases ≤ 2.5 x ULN (in case of liver metastases < 5 x ULN)
* Serum Creatinine ≤ 1.5 x ULN
* Urine dipstick for proteinuria < 2+. If urine dipstick is ≥ 2+, 24- hour urine must demonstrate ≤ 1 g of protein in 24 hours
* Previous adjuvant chemotherapy is allowed if more than 12 months have elapsed between the end of adjuvant therapy and first relapse
* At least 6 weeks from prior radiotherapy and 4 weeks from surgery

Exclusion Criteria:

* Prior palliative chemotherapy
* Prior treatment with bevacizumab
* Bowel obstruction (or subobstruction)
* History of inflammatory enteropathy or extensive intestinal resection (> hemicolectomy or extensive small intestine resection with chronic diarrhea)
* Symptomatic peripheral neuropathy > 2 grade NCIC-CTG criteria
* Presence or history of CNS metastasis
* Active uncontrolled infections
* Active disseminated intravascular coagulation
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to treatment, or anticipation of the need for major surgery during the course of the study
* Central Venous Access Device (CVAD) for chemotherapy administration inserted within 2 days prior to study treatment start
* Past or current history of malignancies other than colorectal carcinoma, except for curatively treated basal and squamous cell carcinoma of the skin cancer or in situ carcinoma of the cervix
* Clinically significant cardiovascular disease, for example cerebrovascular accidents (CVA) (≤ 6 months before treatment start), myocardial infarction (≤ 6 months before treatment start), unstable angina, NYHA ≥ grade 2 chronic heart failure (CHF), uncontrolled arrhythmia
* Uncontrolled hypertension
* 24-hour urine protein > 1 g if dipstick > 2+
* History of thromboembolic or hemorrhagic events within 6 months prior to treatment
* Evidence of bleeding diathesis or coagulopathy
* Serious, non healing wound/ulcer or serious bone fracture
* No therapeutic anticoagulation or antiplatelet agents or NSAID with anti-platelet activity (aspirin ≤ 325 mg/day allowed)
* Pregnancy or lactation
* Fertile women (< 2 years after last menstruation) and men of childbearing potential not willing to use effective means of contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-07; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | PFS rate at 10 months from study entry
  PFS was calculated from the day of treatment start to the first observation of disease progression or death from any cause.

SECONDARY OUTCOMES:
Response rate (RR) | 2007-2010
  Response evaluation was performed every 8 weeks from the day of treatment start until disease progression for each enrolled patient for the full lenght of the study. Response evaluation was performed according to RECIST criteria. Responses were subsequently confirmed by a central review.
Overall survival (OS) | 2007-2010
  OS was calculated from the day of treatment start until death from any cause for each enrolled patient for the full lenght of the study, censoring patients who had not died at the last date known to be alive.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2007-2010
  During the full lenght of first-line treatment, number of enrolled patients reporting adverse events was recorded. Adverse events were evaluated according to National Cancer Institute Common Toxicity Criteria (version 3.0).
Evaluation of potential surrogate markers predictive of bevacizumab activity | 2007-2010
  During first-line therapy and at disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Falcone, MD, Principal Investigator — University of Pisa

REFERENCES:
- [Derived] Cremolini C, Casagrande M, Loupakis F, Aprile G, Bergamo F, Masi G, Moretto R R, Pietrantonio F, Marmorino F, Zucchelli G, Tomasello G, Tonini G, Allegrini G, Granetto C, Ferrari L, Urbani L, Cillo U, Pilati P, Sensi E, Pellegrinelli A, Milione M, Fontanini G, Falcone A. Efficacy of FOLFOXIRI plus bevacizumab in liver-limited metastatic colorectal cancer: A pooled analysis of clinical studies by Gruppo Oncologico del Nord Ovest. Eur J Cancer. 2017 Mar;73:74-84. doi: 10.1016/j.ejca.2016.10.028. Epub 2016 Dec 13. PMID 27986363
- [Derived] Masi G, Loupakis F, Salvatore L, Fornaro L, Cremolini C, Cupini S, Ciarlo A, Del Monte F, Cortesi E, Amoroso D, Granetto C, Fontanini G, Sensi E, Lupi C, Andreuccetti M, Falcone A. Bevacizumab with FOLFOXIRI (irinotecan, oxaliplatin, fluorouracil, and folinate) as first-line treatment for metastatic colorectal cancer: a phase 2 trial. Lancet Oncol. 2010 Sep;11(9):845-52. doi: 10.1016/S1470-2045(10)70175-3. Epub 2010 Aug 9. PMID 20702138